CLINICAL TRIAL: NCT00925860
Title: Non-Positive Pressure Ventilation in Hypoxemic Patients. A Randomized Study
Brief Title: Non-Positive Pressure Ventilation in Hypoxemic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Provincial de Castellon (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGCS-2009-1
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Last update posted 2009-06-22 (Estimated); Status verified 2009-06

CONDITIONS: Acute Respiratory Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- non invasive ventilation approach (Experimental): pure hypoxemic patients admitted to ICU treated by non-positive pressure mechanical ventilation
  Interventions: Procedure: non positive pressure mechanical ventilatory support
- conventionally ventilated (No Intervention): pure hypoxemic patients treated by conventional ventilatory support

INTERVENTIONS:
Procedure: non positive pressure mechanical ventilatory support
  Arms: non invasive ventilation approach

SUMMARY:
The study is aimed to assess the possible benefit of non-positive pressure mechanical support in front of conventional ventilation in patients admitted to the intensive care unit (ICU) because of pure hypoxemic respiratory failure.

DETAILED DESCRIPTION:
Pure hypoxemic patients admitted to intensive care unit in a teaching hospital have been randomized to be treated by conventional ventilatory support or non-positive mechanical ventilation support. Those patients who did not benefit from the experimental non-positive ventilatory support, were intubated and conventionally mechanically ventilated and discarded for analysis. The primary outcome was mortality rate in both groups, and secondary outcomes were length of stay, improvement of oxygenation, and reduced complications rates.

ELIGIBILITY:
Inclusion Criteria:

* dyspnea with respiratory rates higher than 35 p.m.
* pO2 < 65 mmHg
* paO2/FiO2 < 250

Exclusion Criteria:

* respiratory or cardiac arrest
* gastrointestinal bleeding
* hemodynamic instability
* face surgery
* upper airway obstruction
* inability for active cooperation
* need for airway protection
* exacerbation of COPD
* decrease of conscious level
* acute pulmonary cardiogenic oedema

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2001-06; Primary Completion 2006-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
mortality rates | patient hospital discharge

SECONDARY OUTCOMES:
oxygenation improve | patient hospital discharge
diminishing of tracheal intubation incidence | patient hospital discharge
ICU and Post ICU hospital length of stay | patient hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Belenguer, MD, Principal Investigator — INTENSIVE CARE DEPARTMENT, HOSPITAL GENERAL DE CASTELLO
Locations (1):
- Intensive Care Department - General Hospital, Castelló, CASTELLO, Spain